CLINICAL TRIAL: NCT02815748
Title: A Single-center, Randomized, Open, Single Dose Phase I Study to Access the Metabolite Identification and Material Balance in Health Volunteer
Brief Title: The Metabolite Identification and Material Balance Study of SP2086
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-SP2086-109
Record Dates: First submitted 2016-01-03; First posted 2016-06-28 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes
Keywords: SP2086; Metabolite identification; Material balance
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SP2086 (Other): SP2086 was taken only one time at 100mg dose in health volunteers
  Interventions: Drug: SP2086

INTERVENTIONS:
Drug: SP2086 — SP2086 was taken only one time at 100mg dose in health volunteers

SUMMARY:
The purpose of the study is to investigate the Metabolite identification and material balance of SP2086 in healthy adult volunteers.

DETAILED DESCRIPTION:
All subjects were given SP2086 100mg only one time, and blood sample should be collected before and 96 hours after medicine taken.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index(BMI) between 19 and 25 Kg/m2,and weight ≥50kg.
* Lab and other examination results were normal or mildly abnormal without clinical significance, clinical doctors had considered eligible.
* Had signed the informed consent himself or herself voluntarily.

Exclusion Criteria:

* Has a history of severe system disease, or family history (including the cardiovascular system, digestive system, urinary system, etc.).
* Has a history of allergy or intolerance to SP2086 OR other DPP-IV.
* The subjects participated 3 times or more than 3 times drug clinical subjects in nearly a year;participate any drug clinical trial prior to the test 3 months, or had blood donor, or plan to blood donors three months before the test;or had a transfusion in 4 weeks.
* Did not take effective contraceptive measures or planning of the subjects in half a year.
* Researchers considered the patient adherence is poor, or has any unfavorable factors that not suit to participate the test.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SP2086 | up to 96 hours
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of multiple doses of SP2086
The maximum plasma concentration (Cmax) of SP2086 acid | up to 96 hours
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086
The area under the plasma concentration-time curve (AUC) of SP2086 | up to 96 hours
  AUC (a measure of the body's exposure to SP2086) will be compared before and after administration of multiple doses of SP2086
The area under the plasma concentration-time curve (AUC) of SP2086 acid | up to 96 hours
  AUC (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: XingHe Wang, P.H.D, Principal Investigator — Beijing Shijitan Hospital Affiliated to Capital Medical University